CLINICAL TRIAL: NCT03803306
Title: Vedic Medical Astrology in Essential Hypertension: A Double-blind, Placebo-controlled Study
Brief Title: Vedic Medical Astrology in Essential Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (UK) Ltd (Unknown); Swamigal Trust for Vedic Science, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NMP 2172
Record Dates: First submitted 2019-01-11; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vedic Medical Astrology Group (VMA) (Experimental)
  Interventions: Combination Product: Vedic Medical Astrology
- Placebo vedic medical astrology (PMA) (Sham Comparator)
  Interventions: Other: Placebo vedic medical astrology (PMA)

INTERVENTIONS:
Combination Product: Vedic Medical Astrology — Individualised astrological based interventions were given including vedic counselling, diet, colors, gems, mantras and the worship deities as an adjuvent to ongoing conventional treatments
  Arms: Vedic Medical Astrology Group (VMA)
Other: Placebo vedic medical astrology (PMA) — Conventional treatments were followed with counselling and diet suggestions. astrological interventions were not incorporated during the study phase.
  Arms: Placebo vedic medical astrology (PMA)

SUMMARY:
Previous studies have explored the correlation and impact of astrological events in relation of diseases, health concerns and relationship between birth chart and disease risk. Cardiovascular conditions, sleep and fertility were found significantly associated with moon phase. However, to best of our knowledge no study has documented the impact of astrological intervention in disease management.

This is a randomised, multi-center, double blind placebo controlled clinical trial with two parallel arms. This trial aims to evaluate the effectiveness of Vedic medical astrological intervention for patients with mild to moderate hypertension,with respect to decreasing their blood pressure and improving their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 35 and 60 years old, male and female;
* Patients who meet the diagnostic criteria of essential hypertension (
* Patients taking antihypertensive drugs under the supervision of physicians.
* Patients having understanding of our study and willing to comply with astrological protocol.
* Informed consent

Exclusion Criteria:

* Patients who have been diagnosed as secondary hypertension or malignant hypertension
* Patients with comorbid conditions
* Patients with a chronic disease associated or psychiatric conditions which might not suitable for the study
* Patients who had been treated with any other alternative or complementary medicine during the previous three months

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-01-06 (Actual)

PRIMARY OUTCOMES:
Average systolic and average diastolic blood pressure | change from baseline to 12-weeks
  Blood pressure measured by 24-hour ambulatory blood pressure monitoring

SECONDARY OUTCOMES:
Changes in patients Quality of life | change from baseline to 12-weeks
  Health-related quality of life measure by S36

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Study Director — Warwick Research Services (UK) Ltd; Prashanna Chockalingam, Principal Investigator — Warwick Research Services (UK) Ltd; Puneet Sharma, Study Chair — NMP Medical Research Institute, India; Ramanathan Ravisankar, Principal Investigator — Swamigal Trust for Vedic Science, India
Locations (1):
- NMP Medical Reserach Institute, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided